CLINICAL TRIAL: NCT00972192
Title: Effectiveness of Inpatient HIV Voluntary Counseling and Testing in Uganda
Brief Title: Effectiveness of Inpatient Voluntary Counseling and Testing (VCT) in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Prof. Moses Kamya, Makerere University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 23193
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: HIV
Keywords: HIV testing; HIV risk behavior; access to care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inpatient HIV testing (Active Comparator): Participants who were randomized to the intervention group received free HIV testing and counseling immediately after the baseline interview. Patients underwent phlebotomy and serologic testing and results were disclosed the following day with post-test counseling (before they were discharged from the hospital).
  Interventions: Behavioral: Inpatient HIV testing
- HIV testing post-discharge (No Intervention): Participants who were randomized to the control group were given a referral card and an appointment, by the interviewers, to return for free HIV testing and counseling at Mulago hospital one week after discharge. Participants who returned had their transport reimbursed.
  Interventions: Behavioral: Outpatient HIV testing

INTERVENTIONS:
Behavioral: Inpatient HIV testing — Participants who were randomized to the intervention group received free HIV testing and their results before they were discharged from the hospital.
  Other Names: Inpatient VCT
  Arms: Inpatient HIV testing
Behavioral: Outpatient HIV testing — Participants randomised to the control arm received referral for testing post-discharge
  Other Names: Oupatient VCT
  Arms: HIV testing post-discharge

SUMMARY:
This study compared the effectiveness of inpatient routine VCT to referral for post-discharge VCT in terms of the number of new HIV infections identified, linkage to care for HIV infected individuals and reduction in HIV risk behavior.

DETAILED DESCRIPTION:
Ambulatory HIV voluntary testing and counseling (VCT) has become a mainstay of HIV prevention and linkage to care efforts. Despite expansion of these services in sub-Saharan Africa, most individuals admitted for acute illnesses arrive in hospital unaware of their HIV serostatus. Even then, inpatient risk reduction counseling services are not widely available and utilization of HIV testing services in the hospital is rare; most HIV diagnoses are made clinically without the benefit of counseling or antibody testing. The effectiveness of VCT during hospitalization in high-prevalence, resource poor settings has never been formally studied. It has been argued that the circumstances of hospitalization for HIV-associated illness do not allow for the provision of VCT services in this setting: Patients may be too sick to participate meaningfully in risk reduction counseling and the inpatient medical management of acute illness may leave little time for the provision of VCT. There are also several potentially significant differences between ambulatory and inpatient VCT that may limit efficacy in the latter case. First, inpatient counseling during an acute illness may not reduce risk behavior significantly due to competing priorities and messages communicated to patients while in the hospital. Second, HIV risk behavior may already be so infrequent among individuals with complications of advanced HIV disease that there is little margin for further risk reduction. Third, providing VCT during acute hospitalization may not result in effective linkage to existing outpatient follow-up medical care or community-based support services. It may prove very difficult to bridge the gap between the hospital setting and ongoing outpatient care resources. If this is not accomplished, a major goal of the provision of inpatient VCT will be unmet.

This randomized trial compared the impact of free, routine, VCT during hospitalization for acute illness at Mulago Hospital with referral for ambulatory VCT immediately following hospital discharge (which was the current standard of care). We assessed HIV risk behavior and linkage to care outcomes at 3 and 6 months. The following specific aims were addressed:

Aim 1: To determine the number of HIV infections newly identified by offering free VCT routinely to hospitalized patients.

Aim 2: To determine whether routine VCT in hospitalized patients increases partner disclosure and reduces risk behavior at 3 and 6 months.

Aim 3: To determine whether routine VCT in hospitalized patients increases linkage to follow-up HIV care, including available opportunistic infection prophylaxis, antiretroviral treatment, hospice services, and other community-based social services.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Undocumented HIV status
* Fluency in Luganda or English
* Residence within 20 kilometers of Mulago Hospital
* Able to provide informed consent

Exclusion Criteria:

* Patients with altered mental status or who are too ill to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Number of HIV infections newly identified | 6 months

SECONDARY OUTCOMES:
HIV risk behavior and linkage to follow-up HIV care and support | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moses Kamya, MBCHB, Principal Investigator — Makerere University School of Medicine; David Bangsberg, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Background] Wanyenze R, Kamya M, Liechty CA, Ronald A, Guzman DJ, Wabwire-Mangen F, Mayanja-Kizza H, Bangsberg DR. HIV counseling and testing practices at an urban hospital in Kampala, Uganda. AIDS Behav. 2006 Jul;10(4):361-7. doi: 10.1007/s10461-005-9035-9. PMID 16395619